CLINICAL TRIAL: NCT03291743
Title: The Biologic Onset of Crohn's Disease: A Screening Study in First Degree Relatives
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Death of Principal Investigator
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RTDB-2201
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Crohn Disease; Genetic Predisposition; IBD
Keywords: Crohn's; Capsule endoscopy; IBD
MeSH Terms: conditions — Crohn Disease; Genetic Predisposition to Disease | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- First Degree Relative (Experimental): A total of 112 high risk first-degree relatives will be enrolled in total. Patients with Crohn's Disease will be given information about the study when in clinic for routine care to share with their first degree relatives (FDR). Screening will be done using capsule endoscopy.
  Interventions: Device: Capsule endoscopy
- Healthy Controls (Active Comparator): This study will also enroll 35 healthy controls who will be age and sex matched to the first degree relative (FDR) population. Enrollment will begin after 20-25 FDR's have passed screening and will continue at this interval until all controls have been enrolled. Controls will be initially screened by colonoscopy. If enrolled they will undergo capsule endoscopy as well
  Interventions: Device: Capsule endoscopy

INTERVENTIONS:
Device: Capsule endoscopy — PillCam(TM) CROHN'S CAPSULE
  Other Names: PillCam(TM)

SUMMARY:
Pursuing very early diagnosis is standard of care for several diseases including colon cancer, diabetes and liver disease where an early and aggressive diagnostic and therapeutic approach has been shown to change their natural history. Crohn's disease [CD] still lags since commonly at presentation CD has already run a long course, often responding poorly to therapy or requiring surgery. This innovative project proposes a minimally invasive strategy - capsule endoscopy-based screening of first degree relatives [FDR's] of CD patients - to develop tools to diagnose CD at or near its biologic onset.

DETAILED DESCRIPTION:
Crohn's Disease (CD) is a form of inflammatory bowel disease (IBD) that affects the gastrointestinal tract. CD is a chronic, remitting, and relapsing disease that is rarely diagnosed at or near its biological onset. In routine clinical practice, CD diagnosed at the pre-clinical stage is largely by chance during routine screening procedures. Current evidence suggests these earlier diagnoses lead to better treatment outcomes and may even offer clues to better understand the disease's etiology and pathogenesis. Consequently, diagnosing CD at an early stage may offer several advantages including better response to medical treatment; possible avoidance of long term complications and surgery; and long term cost savings.

In the last several years it has become apparent that Crohn's Disease tends to evolve over time from an inflammatory disease to a fibrosing one due to the repeated healing and repair cycles. The fibrosing found in CD is similar to that of other diseases that affect organs like the liver and pancreas. Extensive fibrosis (build-up of excessive scar tissue) does not respond to drug therapy and must be treated with surgery; therefore, surgical intervention (e.g., intestinal resection) is a treatment modality common to CD patients largely due to this indication. Ideally, Crohn's Disease should be diagnosed before this irreversible damage takes place and while the disease is still responsive to medical therapy; however, the disease only comes to medical attention in the presence of symptoms most often associated with severe bowel damage such as obstructions and strictures. Even still, the presence of these symptoms does not always lead to prompt diagnosis. Additionally, this evidence indicates that CD has already run a long course before it becomes symptomatic and further supports the need for earlier diagnosis.

An efficient screening strategy for Crohn's Disease has yet to be identified. To date, colonoscopy is considered the gold-standard as there are no noninvasive tests that can conclusively screen for disease. Screening the general population has been shown to be inefficient due to the overall risk of developing the disease so it is crucial to determine the populations at the greatest risk. Crohn's Disease has proven to have a strong genetic component. Referral center studies published in the last several years have shown that 5-15% of patients with CD have a family history of the disease; therefore, family members of CD patients may constitute an ideal population for screening. Familial studies have focused mostly on first-degree relatives [FDR] and have found that this group is at a higher risk for developing the disease than the general population. In addition, a landmark study published in 2003 showed that >40% of asymptomatic first-degree relatives of CD patients [CD-FDR] had elevated fecal calprotectin-an intestinal inflammation marker that closely reflects disease activity in CD patients-with values between those of healthy controls and FDR's with diagnosed disease. Additional abnormalities such as, Anti-Saccharomyces Cerevisae Antibodies [ASCA] positivity and elevated inflammatory markers-have also been reported in asymptomatic first-degree relatives at a greater proportion than the known risk of developing the disease.

Recently, at another institution, the investigators conducted an ileocolonoscopy-based screening study in 38 first-degree relatives of patients with Crohn's Disease. Identified first-degree relatives were carefully excluded in the presence of digestive symptoms or a medical history that contained possible causes of intestinal inflammation. The healthy control group consisted of 10 age and sex-matched individuals who were scheduled for a colonoscopy due to unrelated reasons (e.g., colon cancer screening or rectal bleeding) and whose results were found to be normal. In both groups, tissue, blood, and stool samples were collected. Median values for fecal calprotectin (FC) and histology were significantly greater in first-degree relatives when compared to the healthy controls. Additionally, colonoscopy identified three different phenotypes within the first-degree relative population: 1) normal, or superimposable to controls; 2) minor lesions (aphthae or small superficial erosions), and 3) typical features of Crohn's Disease. These findings were confirmed with histological scoring that resulted in three highly separated clusters.

That preliminary research supports the idea that screening within this high-risk population allows for earlier diagnosis. Validating these results on a larger scale and with less invasive methods may lead to the development of a screening strategy that can be implemented as part of routine clinical practice. Additionally, more research is needed to further characterize the novel phenotype identified as it may hold crucial clues to the pathogenesis of the disease.

This study seeks to detect asymptomatic, first-degree relatives of patients with established Crohn's Disease in hopes of catching the disease at or near its biologic onset (pre-clinical stage). Screening will be done using the PillCam™ COLON 2 capsule endoscopy system. Capsule findings will be reviewed by Dr. Sorrentino and Dr. Nguyen at the central site. These findings will then be verified using proven ileocolonoscopy methods. Blood, stool, and tissue specimens will be collected for research-related testing and to be stored for further research. Healthy-controls will be enrolled for comparison purposes. The goal of this study is to validate the preliminary data from our pilot study using a multi-center approach.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who are 18-65 years of age
* FDR: Has a first degree relative (mother, father, offspring, or full sibling) who has been diagnosed with Crohn's Disease Healthy Controls: Normal colonoscopy and histology (if applicable) results, and no family history of inflammatory bowel disease (Crohn's Disease and Ulcerative Colitis)
* Willingness to comply with protocol requirements, timelines, and procedures
* Must be able and willing to provide written consent; medical, surgical, and medication history; current and concomitant medication use; and any other documents deemed relevant by the investigator.
* A negative pregnancy test for all female subjects of childbearing potential at the time of consent. Subject must also agree to follow medically approved birth control measures while enrolled

Exclusion Criteria:

* Suspected or confirmed diagnosis of inflammatory bowel disease or any other gastrointestinal disease or condition
* Known medical history of clinically significant cardiovascular, hematologic, orthopedic, rheumatologic, muscular, neurologic (e.g. dementia, seizure disorder, traumatic brain injury), endocrine, ophthalmologic, infectious (e.g. human immunodeficiency virus, tuberculosis, hepatitis), immunologic, renal, pulmonary (e.g. COPD), dermatologic, reproductive, or psychiatric disorders, conditions, or diseases that would present unacceptable risk to study subjects, compromise the acquisition or interpretation of study data, or otherwise interfere with the study subject's participation
* A systolic blood pressure reading ≥ 180 mmHg and/or a diastolic blood pressure reading of ≥ 110 mmHg at screening
* An oral temperature reading of 100.5º F or greater
* Meets any of the following criteria:

  * Use of systemic non-steroidal anti-inflammatory medication (including low-dose aspirin) within 14 days prior to consent
  * History of oral corticosteroid use within 30 days prior to consent
  * Use of IV corticosteroids within 14 days prior to consent
  * Treatment with IV anti-infectives within 30 days prior to consent
  * Treatment with oral anti-infectives within 14 days prior to consent
* Previous or current history of malignancy (including fully excised cutaneous basal cell carcinoma and squamous cell carcinoma)
* History of stem cell or fecal transplant
* History of clinically significant alcoholism or substance abuse in the last 12 months, as defined in the DSM-IV
* Currently has an implanted electrical device (e.g., pacemaker)
* Screening lab results were found to be exclusionary based on the following

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Crohn's Disease in First Degree Relatives by capsule endoscopy screening | coincident at screening
  This study will screen asymptomatic, first-degree relatives of patients with established Crohn's Disease to detect the disease at or near its biologic onset.

SECONDARY OUTCOMES:
Correlation of capsule endoscopy with ileocolonoscopy; characterization of disease state | coincident at screening
  Evaluate the accuracy of capsule endoscopy (CE) in screening for pre-clinical Crohn's Disease by verifying CE findings with ileocolonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Dario R Sorrentino, MD, FRACP, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosnes J, Cattan S, Blain A, Beaugerie L, Carbonnel F, Parc R, Gendre JP. Long-term evolution of disease behavior of Crohn's disease. Inflamm Bowel Dis. 2002 Jul;8(4):244-50. doi: 10.1097/00054725-200207000-00002. PMID 12131607
- [Background] Sorrentino D, Fogel S, Van den Bogaerde J. Surgery for Crohn's disease and anti-TNF agents: the changing scenario. Expert Rev Gastroenterol Hepatol. 2013 Nov;7(8):689-700. doi: 10.1586/17474124.2013.842895. PMID 24161133
- [Background] Danese S, Fiorino G, Fernandes C, Peyrin-Biroulet L. Catching the therapeutic window of opportunity in early Crohn's disease. Curr Drug Targets. 2014;15(11):1056-63. doi: 10.2174/1389450115666140908125738. PMID 25198784
- [Background] Gevers D, Kugathasan S, Denson LA, Vazquez-Baeza Y, Van Treuren W, Ren B, Schwager E, Knights D, Song SJ, Yassour M, Morgan XC, Kostic AD, Luo C, Gonzalez A, McDonald D, Haberman Y, Walters T, Baker S, Rosh J, Stephens M, Heyman M, Markowitz J, Baldassano R, Griffiths A, Sylvester F, Mack D, Kim S, Crandall W, Hyams J, Huttenhower C, Knight R, Xavier RJ. The treatment-naive microbiome in new-onset Crohn's disease. Cell Host Microbe. 2014 Mar 12;15(3):382-392. doi: 10.1016/j.chom.2014.02.005. PMID 24629344
- [Background] Dassopoulos T, Sultan S, Falck-Ytter YT, Inadomi JM, Hanauer SB. American Gastroenterological Association Institute technical review on the use of thiopurines, methotrexate, and anti-TNF-alpha biologic drugs for the induction and maintenance of remission in inflammatory Crohn's disease. Gastroenterology. 2013 Dec;145(6):1464-78.e1-5. doi: 10.1053/j.gastro.2013.10.046. No abstract available. PMID 24267475
- [Background] Cheifetz AS. Management of active Crohn disease. JAMA. 2013 May 22;309(20):2150-8. doi: 10.1001/jama.2013.4466. PMID 23695484
- [Background] D'Haens G, Baert F, van Assche G, Caenepeel P, Vergauwe P, Tuynman H, De Vos M, van Deventer S, Stitt L, Donner A, Vermeire S, Van De Mierop FJ, Coche JR, van der Woude J, Ochsenkuhn T, van Bodegraven AA, Van Hootegem PP, Lambrecht GL, Mana F, Rutgeerts P, Feagan BG, Hommes D; Belgian Inflammatory Bowel Disease Research Group; North-Holland Gut Club. Early combined immunosuppression or conventional management in patients with newly diagnosed Crohn's disease: an open randomised trial. Lancet. 2008 Feb 23;371(9613):660-667. doi: 10.1016/S0140-6736(08)60304-9. PMID 18295023
- [Background] Colombel JF, Sandborn WJ, Rutgeerts P, Enns R, Hanauer SB, Panaccione R, Schreiber S, Byczkowski D, Li J, Kent JD, Pollack PF. Adalimumab for maintenance of clinical response and remission in patients with Crohn's disease: the CHARM trial. Gastroenterology. 2007 Jan;132(1):52-65. doi: 10.1053/j.gastro.2006.11.041. Epub 2006 Nov 29. PMID 17241859
- [Background] Schreiber S, Colombel JF, Bloomfield R, Nikolaus S, Scholmerich J, Panes J, Sandborn WJ; PRECiSE 2 Study Investigators. Increased response and remission rates in short-duration Crohn's disease with subcutaneous certolizumab pegol: an analysis of PRECiSE 2 randomized maintenance trial data. Am J Gastroenterol. 2010 Jul;105(7):1574-82. doi: 10.1038/ajg.2010.78. Epub 2010 Mar 16. PMID 20234346
- [Background] Peyrin-Biroulet L, Bigard MA, Malesci A, Danese S. Step-up and top-down approaches to the treatment of Crohn's disease: early may already be too late. Gastroenterology. 2008 Oct;135(4):1420-2. doi: 10.1053/j.gastro.2008.08.017. Epub 2008 Sep 4. No abstract available. PMID 18773901
- [Background] Rubin DT, Uluscu O, Sederman R. Response to biologic therapy in Crohn's disease is improved with early treatment: an analysis of health claims data. Inflamm Bowel Dis. 2012 Dec;18(12):2225-31. doi: 10.1002/ibd.22925. Epub 2012 Feb 22. PMID 22359399
- [Background] Schoepfer AM, Dehlavi MA, Fournier N, Safroneeva E, Straumann A, Pittet V, Peyrin-Biroulet L, Michetti P, Rogler G, Vavricka SR; IBD Cohort Study Group. Diagnostic delay in Crohn's disease is associated with a complicated disease course and increased operation rate. Am J Gastroenterol. 2013 Nov;108(11):1744-53; quiz 1754. doi: 10.1038/ajg.2013.248. Epub 2013 Aug 27. PMID 23978953
- [Background] Feagan BG, Panaccione R, Sandborn WJ, D'Haens GR, Schreiber S, Rutgeerts PJ, Loftus EV Jr, Lomax KG, Yu AP, Wu EQ, Chao J, Mulani P. Effects of adalimumab therapy on incidence of hospitalization and surgery in Crohn's disease: results from the CHARM study. Gastroenterology. 2008 Nov;135(5):1493-9. doi: 10.1053/j.gastro.2008.07.069. Epub 2008 Aug 3. PMID 18848553
- [Background] Lichtenstein GR, Yan S, Bala M, Blank M, Sands BE. Infliximab maintenance treatment reduces hospitalizations, surgeries, and procedures in fistulizing Crohn's disease. Gastroenterology. 2005 Apr;128(4):862-9. doi: 10.1053/j.gastro.2005.01.048. PMID 15825070
- [Background] Lichtenstein GR, Yan S, Bala M, Hanauer S. Remission in patients with Crohn's disease is associated with improvement in employment and quality of life and a decrease in hospitalizations and surgeries. Am J Gastroenterol. 2004 Jan;99(1):91-6. doi: 10.1046/j.1572-0241.2003.04010.x. PMID 14687148
- [Background] Leombruno JP, Nguyen GC, Grootendorst P, Juurlink D, Einarson T. Hospitalization and surgical rates in patients with Crohn's disease treated with infliximab: a matched analysis. Pharmacoepidemiol Drug Saf. 2011 Aug;20(8):838-48. doi: 10.1002/pds.2132. Epub 2011 Jun 17. PMID 21688345
- [Background] Benevento G, Avellini C, Terrosu G, Geraci M, Lodolo I, Sorrentino D. Diagnosis and assessment of Crohn's disease: the present and the future. Expert Rev Gastroenterol Hepatol. 2010 Dec;4(6):757-66. doi: 10.1586/egh.10.70. PMID 21108595
- [Background] Vavricka SR, Spigaglia SM, Rogler G, Pittet V, Michetti P, Felley C, Mottet C, Braegger CP, Rogler D, Straumann A, Bauerfeind P, Fried M, Schoepfer AM; Swiss IBD Cohort Study Group. Systematic evaluation of risk factors for diagnostic delay in inflammatory bowel disease. Inflamm Bowel Dis. 2012 Mar;18(3):496-505. doi: 10.1002/ibd.21719. Epub 2011 Apr 20. PMID 21509908
- [Background] Hovde O, Moum BA. Epidemiology and clinical course of Crohn's disease: results from observational studies. World J Gastroenterol. 2012 Apr 21;18(15):1723-31. doi: 10.3748/wjg.v18.i15.1723. PMID 22553396
- [Background] Burgmann T, Clara I, Graff L, Walker J, Lix L, Rawsthorne P, McPhail C, Rogala L, Miller N, Bernstein CN. The Manitoba Inflammatory Bowel Disease Cohort Study: prolonged symptoms before diagnosis--how much is irritable bowel syndrome? Clin Gastroenterol Hepatol. 2006 May;4(5):614-20. doi: 10.1016/j.cgh.2006.03.003. Epub 2006 Apr 17. PMID 16630762
- [Background] Thjodleifsson B, Sigthorsson G, Cariglia N, Reynisdottir I, Gudbjartsson DF, Kristjansson K, Meddings JB, Gudnason V, Wandall JH, Andersen LP, Sherwood R, Kjeld M, Oddsson E, Gudjonsson H, Bjarnason I. Subclinical intestinal inflammation: an inherited abnormality in Crohn's disease relatives? Gastroenterology. 2003 Jun;124(7):1728-37. doi: 10.1016/s0016-5085(03)00383-4. PMID 12806605
- [Background] Sorrentino D, Avellini C, Geraci M, Dassopoulos T, Zarifi D, Vadala' di Prampero SF, Benevento G. Tissue studies in screened first-degree relatives reveal a distinct Crohn's disease phenotype. Inflamm Bowel Dis. 2014 Jun;20(6):1049-56. doi: 10.1097/MIB.0000000000000051. PMID 24788221
- [Background] Sorrentino D. Role of biologics and other therapies in stricturing Crohn's disease: what have we learnt so far? Digestion. 2008;77(1):38-47. doi: 10.1159/000117306. Epub 2008 Feb 19. PMID 18285676
- [Background] Mayberry JF, Ballantyne KC, Hardcastle JD, Mangham C, Pye G. Epidemiological study of asymptomatic inflammatory bowel disease: the identification of cases during a screening programme for colorectal cancer. Gut. 1989 Apr;30(4):481-3. doi: 10.1136/gut.30.4.481. PMID 2785474
- [Background] Sorrentino D. Preclinical and Undiagnosed Crohn's Disease: The Submerged Iceberg. Inflamm Bowel Dis. 2016 Feb;22(2):476-86. doi: 10.1097/MIB.0000000000000612. PMID 26752471
- [Background] Harris R, Sawaya GF, Moyer VA, Calonge N. Reconsidering the criteria for evaluating proposed screening programs: reflections from 4 current and former members of the U.S. Preventive services task force. Epidemiol Rev. 2011;33:20-35. doi: 10.1093/epirev/mxr005. Epub 2011 Jun 10. PMID 21666224
- [Background] Geboes K. The strategy for biopsies of the terminal ileum should be evidence based. Am J Gastroenterol. 2007 May;102(5):1090-2. doi: 10.1111/j.1572-0241.2007.01190.x. PMID 17489785
- [Background] Fries W, Renda MC, Lo Presti MA, Raso A, Orlando A, Oliva L, Giofre MR, Maggio A, Mattaliano A, Macaluso A, Cottone M. Intestinal permeability and genetic determinants in patients, first-degree relatives, and controls in a high-incidence area of Crohn's disease in Southern Italy. Am J Gastroenterol. 2005 Dec;100(12):2730-6. doi: 10.1111/j.1572-0241.2005.00325.x. PMID 16393227
- [Background] Orholm M, Fonager K, Sorensen HT. Risk of ulcerative colitis and Crohn's disease among offspring of patients with chronic inflammatory bowel disease. Am J Gastroenterol. 1999 Nov;94(11):3236-8. doi: 10.1111/j.1572-0241.1999.01526.x. PMID 10566721
- [Background] Ahmad T, Satsangi J, McGovern D, Bunce M, Jewell DP. Review article: the genetics of inflammatory bowel disease. Aliment Pharmacol Ther. 2001 Jun;15(6):731-48. doi: 10.1046/j.1365-2036.2001.00981.x. PMID 11380312
- [Background] Pham M, Leach ST, Lemberg DA, Day AS. Subclinical intestinal inflammation in siblings of children with Crohn's disease. Dig Dis Sci. 2010 Dec;55(12):3502-7. doi: 10.1007/s10620-010-1434-8. Epub 2010 Oct 8. PMID 20931283
- [Background] Montalto M, Curigliano V, Santoro L, Armuzzi A, Cammarota G, Covino M, Mentella MC, Ancarani F, Manna R, Gasbarrini A, Gasbarrini G. Fecal calprotectin in first-degree relatives of patients with ulcerative colitis. Am J Gastroenterol. 2007 Jan;102(1):132-6. doi: 10.1111/j.1572-0241.2006.00884.x. Epub 2006 Nov 13. PMID 17100982
- [Background] Tamboli CP, Richard F, Colombel JF. Fecal calprotectin in Crohn's disease: new family ties. Gastroenterology. 2003 Jun;124(7):1972-4. doi: 10.1016/s0016-5085(03)00552-3. No abstract available. PMID 12806631
- [Background] Soderholm JD, Olaison G, Lindberg E, Hannestad U, Vindels A, Tysk C, Jarnerot G, Sjodahl R. Different intestinal permeability patterns in relatives and spouses of patients with Crohn's disease: an inherited defect in mucosal defence? Gut. 1999 Jan;44(1):96-100. doi: 10.1136/gut.44.1.96. PMID 9862833
- [Background] Sendid B, Quinton JF, Charrier G, Goulet O, Cortot A, Grandbastien B, Poulain D, Colombel JF. Anti-Saccharomyces cerevisiae mannan antibodies in familial Crohn's disease. Am J Gastroenterol. 1998 Aug;93(8):1306-10. doi: 10.1111/j.1572-0241.1998.00415.x. PMID 9707056
- [Background] Ananthakrishnan AN. Environmental risk factors for inflammatory bowel diseases: a review. Dig Dis Sci. 2015 Feb;60(2):290-8. doi: 10.1007/s10620-014-3350-9. Epub 2014 Sep 10. PMID 25204669
- [Background] Peeters M, Geypens B, Claus D, Nevens H, Ghoos Y, Verbeke G, Baert F, Vermeire S, Vlietinck R, Rutgeerts P. Clustering of increased small intestinal permeability in families with Crohn's disease. Gastroenterology. 1997 Sep;113(3):802-7. doi: 10.1016/s0016-5085(97)70174-4. PMID 9287971
- [Background] Israeli E, Grotto I, Gilburd B, Balicer RD, Goldin E, Wiik A, Shoenfeld Y. Anti-Saccharomyces cerevisiae and antineutrophil cytoplasmic antibodies as predictors of inflammatory bowel disease. Gut. 2005 Sep;54(9):1232-6. doi: 10.1136/gut.2004.060228. PMID 16099791
- [Background] Efrat B, Iris G, Wang H, Eitan S, Yona K. A subgroup of first-degree relatives of Crohn's disease patients shows a profile of inflammatory markers in the blood which is more typical of Crohn's disease patients than of normal individuals. Mediators Inflamm. 2006;2006(2):74785. doi: 10.1155/MI/2006/74785. PMID 16883067
- [Background] Annese V, Andreoli A, Andriulli A, Dinca R, Gionchetti P, Latiano A, Lombardi G, Piepoli A, Poulain D, Sendid B, Colombel JF. Familial expression of anti-Saccharomyces cerevisiae Mannan antibodies in Crohn's disease and ulcerative colitis: a GISC study. Am J Gastroenterol. 2001 Aug;96(8):2407-12. doi: 10.1111/j.1572-0241.2001.04043.x. PMID 11513182
- [Background] Elmgreen J, Both H, Binder V. Familial occurrence of complement dysfunction in Crohn's disease: correlation with intestinal symptoms and hypercatabolism of complement. Gut. 1985 Feb;26(2):151-7. doi: 10.1136/gut.26.2.151. PMID 3967833
- [Background] Joossens M, Huys G, Cnockaert M, De Preter V, Verbeke K, Rutgeerts P, Vandamme P, Vermeire S. Dysbiosis of the faecal microbiota in patients with Crohn's disease and their unaffected relatives. Gut. 2011 May;60(5):631-7. doi: 10.1136/gut.2010.223263. Epub 2011 Jan 5. PMID 21209126
- [Background] Mei L, Targan SR, Landers CJ, Dutridge D, Ippoliti A, Vasiliauskas EA, Papadakis KA, Fleshner PR, Rotter JI, Yang H. Familial expression of anti-Escherichia coli outer membrane porin C in relatives of patients with Crohn's disease. Gastroenterology. 2006 Apr;130(4):1078-85. doi: 10.1053/j.gastro.2006.02.013. PMID 16618402
- [Background] Devlin SM, Yang H, Ippoliti A, Taylor KD, Landers CJ, Su X, Abreu MT, Papadakis KA, Vasiliauskas EA, Melmed GY, Fleshner PR, Mei L, Rotter JI, Targan SR. NOD2 variants and antibody response to microbial antigens in Crohn's disease patients and their unaffected relatives. Gastroenterology. 2007 Feb;132(2):576-86. doi: 10.1053/j.gastro.2006.11.013. Epub 2006 Nov 10. PMID 17258734
- [Background] Folwaczny C, Noehl N, Endres SP, Heldwein W, Loeschke K, Fricke H. Antinuclear autoantibodies in patients with inflammatory bowel disease. High prevalence in first-degree relatives. Dig Dis Sci. 1997 Aug;42(8):1593-7. doi: 10.1023/a:1018832608899. PMID 9286222
- [Background] Folwaczny C, Noehl N, Tschop K, Endres SP, Heldwein W, Loeschke K, Fricke H. Goblet cell autoantibodies in patients with inflammatory bowel disease and their first-degree relatives. Gastroenterology. 1997 Jul;113(1):101-6. doi: 10.1016/s0016-5085(97)70085-4. PMID 9207267
- [Background] Bjarnason I, Helgason KO, Geirsson AJ, Sigthorsson G, Reynisdottir I, Gudbjartsson D, Einarsdottir AS, Sherwood R, Kristjansson K, Kjartansson O, Thjodleifsson B. Subclinical intestinal inflammation and sacroiliac changes in relatives of patients with ankylosing spondylitis. Gastroenterology. 2003 Dec;125(6):1598-605. doi: 10.1053/j.gastro.2003.08.035. PMID 14724811
- [Background] Dorn SD, Abad JF, Panagopoulos G, Korelitz BI. Clinical characteristics of familial versus sporadic Crohn's disease using the Vienna Classification. Inflamm Bowel Dis. 2004 May;10(3):201-6. doi: 10.1097/00054725-200405000-00004. PMID 15290912
- [Background] D'Haens GR, Geboes K, Peeters M, Baert F, Penninckx F, Rutgeerts P. Early lesions of recurrent Crohn's disease caused by infusion of intestinal contents in excluded ileum. Gastroenterology. 1998 Feb;114(2):262-7. doi: 10.1016/s0016-5085(98)70476-7. PMID 9453485
- [Background] Sandborn WJ, Feagan BG, Hanauer SB, Lochs H, Lofberg R, Modigliani R, Present DH, Rutgeerts P, Scholmerich J, Stange EF, Sutherland LR. A review of activity indices and efficacy endpoints for clinical trials of medical therapy in adults with Crohn's disease. Gastroenterology. 2002 Feb;122(2):512-30. doi: 10.1053/gast.2002.31072. No abstract available. PMID 11832465
- [Background] Zwas FR, Cirillo NW, el-Serag HB, Eisen RN. Colonic mucosal abnormalities associated with oral sodium phosphate solution. Gastrointest Endosc. 1996 May;43(5):463-6. doi: 10.1016/s0016-5107(96)70286-9. PMID 8726758
- [Background] Zhulina Y, Hahn-Stromberg V, Shamikh A, Peterson CG, Gustavsson A, Nyhlin N, Wickbom A, Bohr J, Bodin L, Tysk C, Carlson M, Halfvarson J. Subclinical inflammation with increased neutrophil activity in healthy twin siblings reflect environmental influence in the pathogenesis of inflammatory bowel disease. Inflamm Bowel Dis. 2013 Jul;19(8):1725-31. doi: 10.1097/MIB.0b013e318281f2d3. PMID 23669399
- [Background] Krauss E, Agaimy A, Neumann H, Schulz U, Kessler H, Hartmann A, Neurath MF, Raithel M, Mudter J. Characterization of lymphoid follicles with red ring signs as first manifestation of early Crohn's disease by conventional histopathology and confocal laser endomicroscopy. Int J Clin Exp Pathol. 2012;5(5):411-21. Epub 2012 May 23. PMID 22808293
- [Background] Fujimura Y, Kamoi R, Iida M. Pathogenesis of aphthoid ulcers in Crohn's disease: correlative findings by magnifying colonoscopy, electron microscopy, and immunohistochemistry. Gut. 1996 May;38(5):724-32. doi: 10.1136/gut.38.5.724. PMID 8707119
- [Background] Gullberg E, Soderholm JD. Peyer's patches and M cells as potential sites of the inflammatory onset in Crohn's disease. Ann N Y Acad Sci. 2006 Aug;1072:218-32. doi: 10.1196/annals.1326.028. PMID 17057202
- [Background] Morson BC. The early histological lesion of Crohn's disease. Proc R Soc Med. 1972 Jan;65(1):71-2. doi: 10.1177/003591577206500129. No abstract available. PMID 5015484
- [Background] Maloy KJ, Powrie F. Intestinal homeostasis and its breakdown in inflammatory bowel disease. Nature. 2011 Jun 15;474(7351):298-306. doi: 10.1038/nature10208. PMID 21677746
- [Background] Zorzi F, Monteleone I, Sarra M, Calabrese E, Marafini I, Cretella M, Sedda S, Biancone L, Pallone F, Monteleone G. Distinct profiles of effector cytokines mark the different phases of Crohn's disease. PLoS One. 2013;8(1):e54562. doi: 10.1371/journal.pone.0054562. Epub 2013 Jan 17. PMID 23349929
- [Background] Hedin CR, McCarthy NE, Louis P, Farquharson FM, McCartney S, Taylor K, Prescott NJ, Murrells T, Stagg AJ, Whelan K, Lindsay JO. Altered intestinal microbiota and blood T cell phenotype are shared by patients with Crohn's disease and their unaffected siblings. Gut. 2014 Oct;63(10):1578-86. doi: 10.1136/gutjnl-2013-306226. Epub 2014 Jan 7. PMID 24398881
- [Background] Kostic AD, Xavier RJ, Gevers D. The microbiome in inflammatory bowel disease: current status and the future ahead. Gastroenterology. 2014 May;146(6):1489-99. doi: 10.1053/j.gastro.2014.02.009. Epub 2014 Feb 19. PMID 24560869
- [Background] Sartor RB. Genetics and environmental interactions shape the intestinal microbiome to promote inflammatory bowel disease versus mucosal homeostasis. Gastroenterology. 2010 Dec;139(6):1816-9. doi: 10.1053/j.gastro.2010.10.036. Epub 2010 Oct 26. No abstract available. PMID 21029802
- [Background] Mukherjee PK, Sendid B, Hoarau G, Colombel JF, Poulain D, Ghannoum MA. Mycobiota in gastrointestinal diseases. Nat Rev Gastroenterol Hepatol. 2015 Feb;12(2):77-87. doi: 10.1038/nrgastro.2014.188. Epub 2014 Nov 11. PMID 25385227
- [Background] Moyes DL, Naglik JR. The mycobiome: influencing IBD severity. Cell Host Microbe. 2012 Jun 14;11(6):551-2. doi: 10.1016/j.chom.2012.05.009. PMID 22704612
- [Background] Iliev ID, Funari VA, Taylor KD, Nguyen Q, Reyes CN, Strom SP, Brown J, Becker CA, Fleshner PR, Dubinsky M, Rotter JI, Wang HL, McGovern DP, Brown GD, Underhill DM. Interactions between commensal fungi and the C-type lectin receptor Dectin-1 influence colitis. Science. 2012 Jun 8;336(6086):1314-7. doi: 10.1126/science.1221789. Epub 2012 Jun 6. PMID 22674328
- [Background] Standaert-Vitse A, Sendid B, Joossens M, Francois N, Vandewalle-El Khoury P, Branche J, Van Kruiningen H, Jouault T, Rutgeerts P, Gower-Rousseau C, Libersa C, Neut C, Broly F, Chamaillard M, Vermeire S, Poulain D, Colombel JF. Candida albicans colonization and ASCA in familial Crohn's disease. Am J Gastroenterol. 2009 Jul;104(7):1745-53. doi: 10.1038/ajg.2009.225. Epub 2009 May 26. PMID 19471251
- [Background] Hedin CR, Stagg AJ, Whelan K, Lindsay JO. Family studies in Crohn's disease: new horizons in understanding disease pathogenesis, risk and prevention. Gut. 2012 Feb;61(2):311-8. doi: 10.1136/gut.2011.238568. Epub 2011 May 11. PMID 21561876
- [Background] Sorrentino D, Avellini C, Geraci M, Vadala S. Pre-clinical Crohn's disease: diagnosis, treatment and six year follow-up. J Crohns Colitis. 2014 Jul;8(7):702-7. doi: 10.1016/j.crohns.2013.12.008. Epub 2014 Jan 8. PMID 24411923
- [Background] Barnes MJ, Powrie F. Regulatory T cells reinforce intestinal homeostasis. Immunity. 2009 Sep 18;31(3):401-11. doi: 10.1016/j.immuni.2009.08.011. PMID 19766083
- [Background] Fantini MC, Rizzo A, Fina D, Caruso R, Sarra M, Stolfi C, Becker C, Macdonald TT, Pallone F, Neurath MF, Monteleone G. Smad7 controls resistance of colitogenic T cells to regulatory T cell-mediated suppression. Gastroenterology. 2009 Apr;136(4):1308-16, e1-3. doi: 10.1053/j.gastro.2008.12.053. Epub 2008 Dec 27. PMID 19192480
- [Background] Strober W, Fuss IJ. Proinflammatory cytokines in the pathogenesis of inflammatory bowel diseases. Gastroenterology. 2011 May;140(6):1756-1767. doi: 10.1053/j.gastro.2011.02.016. PMID 21530742
- [Background] Papp M, Lakatos PL. Serological studies in inflammatory bowel disease: how important are they? Curr Opin Gastroenterol. 2014 Jul;30(4):359-64. doi: 10.1097/MOG.0000000000000076. PMID 24811052
- [Background] van Schaik FD, Oldenburg B, Hart AR, Siersema PD, Lindgren S, Grip O, Teucher B, Kaaks R, Bergmann MM, Boeing H, Carbonnel F, Jantchou P, Boutron-Ruault MC, Tjonneland A, Olsen A, Crowe FL, Peeters PH, van Oijen MG, Bueno-de-Mesquita HB. Serological markers predict inflammatory bowel disease years before the diagnosis. Gut. 2013 May;62(5):683-8. doi: 10.1136/gutjnl-2012-302717. Epub 2012 Jul 26. PMID 22842615
- [Background] Lonnkvist MH, Theodorsson E, Holst M, Ljung T, Hellstrom PM. Blood chemistry markers for evaluation of inflammatory activity in Crohn's disease during infliximab therapy. Scand J Gastroenterol. 2011 Apr;46(4):420-7. doi: 10.3109/00365521.2010.539253. Epub 2010 Nov 30. PMID 21114432
- [Background] Kopylov U, Rosenfeld G, Bressler B, Seidman E. Clinical utility of fecal biomarkers for the diagnosis and management of inflammatory bowel disease. Inflamm Bowel Dis. 2014 Apr;20(4):742-56. doi: 10.1097/01.MIB.0000442681.85545.31. PMID 24562174
- [Background] Sorrentino D, Terrosu G, Paviotti A, Geraci M, Avellini C, Zoli G, Fries W, Danese S, Occhipinti P, Croatto T, Zarifi D. Early diagnosis and treatment of postoperative endoscopic recurrence of Crohn's disease: partial benefit by infliximab--a pilot study. Dig Dis Sci. 2012 May;57(5):1341-8. doi: 10.1007/s10620-011-2025-z. Epub 2012 Jan 18. PMID 22252267
- [Background] Sorrentino D, Paviotti A, Terrosu G, Avellini C, Geraci M, Zarifi D. Low-dose maintenance therapy with infliximab prevents postsurgical recurrence of Crohn's disease. Clin Gastroenterol Hepatol. 2010 Jul;8(7):591-9.e1; quiz e78-9. doi: 10.1016/j.cgh.2010.01.016. Epub 2010 Feb 4. PMID 20139033
- [Background] Hyams J, Crandall W, Kugathasan S, Griffiths A, Olson A, Johanns J, Liu G, Travers S, Heuschkel R, Markowitz J, Cohen S, Winter H, Veereman-Wauters G, Ferry G, Baldassano R; REACH Study Group. Induction and maintenance infliximab therapy for the treatment of moderate-to-severe Crohn's disease in children. Gastroenterology. 2007 Mar;132(3):863-73; quiz 1165-6. doi: 10.1053/j.gastro.2006.12.003. Epub 2006 Dec 3. PMID 17324398
- [Background] Goutorbe F, Goutte M, Minet-Quinard R, Boucher AL, Pereira B, Bommelaer G, Buisson A. Endoscopic Factors Influencing Fecal Calprotectin Value in Crohn's Disease. J Crohns Colitis. 2015 Dec;9(12):1113-9. doi: 10.1093/ecco-jcc/jjv150. Epub 2015 Sep 7. PMID 26351383
- [Background] Sipponen T, Karkkainen P, Savilahti E, Kolho KL, Nuutinen H, Turunen U, Farkkila M. Correlation of faecal calprotectin and lactoferrin with an endoscopic score for Crohn's disease and histological findings. Aliment Pharmacol Ther. 2008 Nov 15;28(10):1221-9. doi: 10.1111/j.1365-2036.2008.03835.x. Epub 2008 Aug 26. PMID 18752630
- [Background] Soubieres AA, Poullis A. Emerging role of novel biomarkers in the diagnosis of inflammatory bowel disease. World J Gastrointest Pharmacol Ther. 2016 Feb 6;7(1):41-50. doi: 10.4292/wjgpt.v7.i1.41. PMID 26855811
- [Background] Albert JG, Kotsch J, Kostler W, Behl S, Kaltz B, Bokemeyer B, Dollinger MM, Haerting J, Fleig WE. Course of Crohn's disease prior to establishment of the diagnosis. Z Gastroenterol. 2008 Feb;46(2):187-92. doi: 10.1055/s-2007-963524. PMID 18253897
- [Background] Li Y, Ren J, Wang G, Gu G, Wu X, Ren H, Hong Z, Hu D, Wu Q, Li G, Liu S, Anjum N, Li J. Diagnostic delay in Crohn's disease is associated with increased rate of abdominal surgery: A retrospective study in Chinese patients. Dig Liver Dis. 2015 Jul;47(7):544-8. doi: 10.1016/j.dld.2015.03.004. Epub 2015 Mar 14. PMID 25840874
- [Background] Pellino G, Sciaudone G, Selvaggi F, Riegler G. Delayed diagnosis is influenced by the clinical pattern of Crohn's disease and affects treatment outcomes and quality of life in the long term: a cross-sectional study of 361 patients in Southern Italy. Eur J Gastroenterol Hepatol. 2015 Feb;27(2):175-81. doi: 10.1097/MEG.0000000000000244. PMID 25461228
- [Background] Louis E, Collard A, Oger AF, Degroote E, Aboul Nasr El Yafi FA, Belaiche J. Behaviour of Crohn's disease according to the Vienna classification: changing pattern over the course of the disease. Gut. 2001 Dec;49(6):777-82. doi: 10.1136/gut.49.6.777. PMID 11709511
- [Background] Solberg IC, Vatn MH, Hoie O, Stray N, Sauar J, Jahnsen J, Moum B, Lygren I; IBSEN Study Group. Clinical course in Crohn's disease: results of a Norwegian population-based ten-year follow-up study. Clin Gastroenterol Hepatol. 2007 Dec;5(12):1430-8. doi: 10.1016/j.cgh.2007.09.002. PMID 18054751
- [Background] Kelly JK, Sutherland LR. The chronological sequence in the pathology of Crohn's disease. J Clin Gastroenterol. 1988 Feb;10(1):28-33. doi: 10.1097/00004836-198802000-00008. PMID 3356881
- [Background] Greenstein AJ, Lachman P, Sachar DB, Springhorn J, Heimann T, Janowitz HD, Aufses AH Jr. Perforating and non-perforating indications for repeated operations in Crohn's disease: evidence for two clinical forms. Gut. 1988 May;29(5):588-92. doi: 10.1136/gut.29.5.588. PMID 3396946
- [Background] Limketkai BN, Bayless TM. Editorial: Can stenosis in ileal Crohn's disease be prevented by current therapy? Am J Gastroenterol. 2013 Nov;108(11):1755-6. doi: 10.1038/ajg.2013.301. PMID 24192948
- [Background] Jacene HA, Ginsburg P, Kwon J, Nguyen GC, Montgomery EA, Bayless TM, Wahl RL. Prediction of the need for surgical intervention in obstructive Crohn's disease by 18F-FDG PET/CT. J Nucl Med. 2009 Nov;50(11):1751-9. doi: 10.2967/jnumed.109.065466. Epub 2009 Oct 16. PMID 19837758
- [Background] Cummings SA, Rubin DT. The complexity and challenges of genetic counseling and testing for inflammatory bowel disease. J Genet Couns. 2006 Dec;15(6):465-76. doi: 10.1007/s10897-006-9057-0. PMID 17106630
- [Background] Liu JZ, Anderson CA. Genetic studies of Crohn's disease: past, present and future. Best Pract Res Clin Gastroenterol. 2014 Jun;28(3):373-86. doi: 10.1016/j.bpg.2014.04.009. Epub 2014 May 6. PMID 24913378
- [Background] Leighton JA, Gralnek IM, Cohen SA, Toth E, Cave DR, Wolf DC, Mullin GE, Ketover SR, Legnani PE, Seidman EG, Crowell MD, Bergwerk AJ, Peled R, Eliakim R. Capsule endoscopy is superior to small-bowel follow-through and equivalent to ileocolonoscopy in suspected Crohn's disease. Clin Gastroenterol Hepatol. 2014 Apr;12(4):609-15. doi: 10.1016/j.cgh.2013.09.028. Epub 2013 Sep 27. PMID 24075891
- [Background] Triester SL, Leighton JA, Leontiadis GI, Gurudu SR, Fleischer DE, Hara AK, Heigh RI, Shiff AD, Sharma VK. A meta-analysis of the yield of capsule endoscopy compared to other diagnostic modalities in patients with non-stricturing small bowel Crohn's disease. Am J Gastroenterol. 2006 May;101(5):954-64. doi: 10.1111/j.1572-0241.2006.00506.x. PMID 16696781
- [Background] Jensen MD, Nathan T, Rafaelsen SR, Kjeldsen J. Diagnostic accuracy of capsule endoscopy for small bowel Crohn's disease is superior to that of MR enterography or CT enterography. Clin Gastroenterol Hepatol. 2011 Feb;9(2):124-9. doi: 10.1016/j.cgh.2010.10.019. Epub 2010 Nov 5. PMID 21056692
- [Background] Sipponen T, Haapamaki J, Savilahti E, Alfthan H, Hamalainen E, Rautiainen H, Koskenpato J, Nuutinen H, Farkkila M. Fecal calprotectin and S100A12 have low utility in prediction of small bowel Crohn's disease detected by wireless capsule endoscopy. Scand J Gastroenterol. 2012 Jul;47(7):778-84. doi: 10.3109/00365521.2012.677953. Epub 2012 Apr 23. PMID 22519419
- [Background] Maiden L, Thjodleifsson B, Theodors A, Gonzalez J, Bjarnason I. A quantitative analysis of NSAID-induced small bowel pathology by capsule enteroscopy. Gastroenterology. 2005 May;128(5):1172-8. doi: 10.1053/j.gastro.2005.03.020. PMID 15887101
- [Background] Gralnek IM, Defranchis R, Seidman E, Leighton JA, Legnani P, Lewis BS. Development of a capsule endoscopy scoring index for small bowel mucosal inflammatory change. Aliment Pharmacol Ther. 2008 Jan 15;27(2):146-54. doi: 10.1111/j.1365-2036.2007.03556.x. Epub 2007 Oct 23. PMID 17956598
- [Background] Biancone L, Calabrese E, Petruzziello C, Capanna A, Zorzi F, Onali S, Condino G, Lolli E, Ciccacci C, Borgiani P, Pallone F. A family study of asymptomatic small bowel Crohn's disease. Dig Liver Dis. 2014 Mar;46(3):276-8. doi: 10.1016/j.dld.2013.11.003. Epub 2013 Dec 17. PMID 24360029
- [Background] Sands BE. From symptom to diagnosis: clinical distinctions among various forms of intestinal inflammation. Gastroenterology. 2004 May;126(6):1518-32. doi: 10.1053/j.gastro.2004.02.072. No abstract available. PMID 15168364
- [Background] Bennett RA, Rubin PH, Present DH. Frequency of inflammatory bowel disease in offspring of couples both presenting with inflammatory bowel disease. Gastroenterology. 1991 Jun;100(6):1638-43. doi: 10.1016/0016-5085(91)90663-6. PMID 2019369
- [Background] Noble CL, Arnott ID. What is the risk that a child will develop inflammatory bowel disease if 1 or both parents have IBD? Inflamm Bowel Dis. 2008 Oct;14 Suppl 2:S22-3. doi: 10.1002/ibd.20575. No abstract available. PMID 18816708
- [Background] Russell RK, Satsangi J. Does IBD run in families? Inflamm Bowel Dis. 2008 Oct;14 Suppl 2:S20-1. doi: 10.1002/ibd.20573. No abstract available. PMID 18816757
- [Background] Probert CS, Brown M. Are there any ethnic groups that are more likely to develop IBD? Inflamm Bowel Dis. 2008 Oct;14 Suppl 2:S24-5. doi: 10.1002/ibd.20601. No abstract available. PMID 18816723
- [Background] Yan B, Panaccione R, Sutherland L. I am Jewish: what is my risk of developing Crohn's disease? Inflamm Bowel Dis. 2008 Oct;14 Suppl 2:S26-7. doi: 10.1002/ibd.20691. No abstract available. PMID 18816782
- [Background] Shrout PE, Fleiss JL. Intraclass correlations: uses in assessing rater reliability. Psychol Bull. 1979 Mar;86(2):420-8. doi: 10.1037//0033-2909.86.2.420. PMID 18839484